CLINICAL TRIAL: NCT01817647
Title: PREDICS Study: Procalcitonin Reveals Early Dehiscence in Colorectal Surgery
Brief Title: PREDICS Study: PCT Reveals Early Dehiscence in Colorectal Surgery
Acronym: PREDICS
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Valentina Giaccaglia, MD, University of Roma La Sapienza
Other Study IDs: PCT-2013
Record Dates: First submitted 2013-03-20; First posted 2013-03-25 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Anastomotic Leak
Keywords: AL; Enhanced recovery after surgery (ERAS); reduce postoperative complications; increased risk of delayed diagnosis and treatment of AL; diagnose anastomotic leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCT: Patients undergoing colorectal surgery with an anastomosis performed
  Interventions: Procedure: Colorectal surgery

INTERVENTIONS:
Procedure: Colorectal surgery

SUMMARY:
Procalcitonin (PCT) is a biomarker used to monitor serious bacterial infections and guide antibiotic therapy. Anastomotic leak (AL) after colorectal surgery is a severe complication associated with relevant short and long-term sequelae. The aim of our study is to assess the predictive value of PCT level for early diagnosis of anastomotic leak after colorectal surgery.

DETAILED DESCRIPTION:
Anastomotic leak (AL) after colorectal surgery represents a major clinical problem observed in a range from 2 to 7% of patients, rising up to 14% in low colorectal resections, and even to 26% in some older reports.1-3 Enhanced recovery after surgery (ERAS) programs are nowadays proven to reduce postoperative complications in up to 50% of cases, fasten recovery and shorten length of stay.4-5 These fast-track protocols demand very early patient discharge but this might be potentially associated with an increased risk of delayed diagnosis and treatment of AL occurring after patient discharge. Hence, there is a strong need of an additional tool to early diagnose anastomotic leak, prior patient discharge. Serum procalcitonin (PCT), is a 116 amino-acids protein produced by C-cells of the thyroid gland. PCT baseline levels are low (<0.1 ng/ml), but increase significantly in patients with severe bacterial infections. Therefore, PCT levels are used to monitor the course and prognosis of systemic bacterial infections and to tailor the therapeutic interventions more efficiently.6-7 Furthermore, PCT could serve as an early predictive marker for the clinical course of septic complications after abdominal surgery.8-9 The aim of our study is to demonstrate if PCT is a more sensible, specific and reliable biomarker of anastomotic leak (AL) than CRP and WBC and if PCT is < 5 ng/ml in 5th POD might be safely added as an additional criteria of early discharge in ERAS protocols.

All patients undergoing colorectal surgery in our centre, either electively or in emergency setting, are recruited. In all cases white blood count (WBC), C-reactive protein (CRP) and PCT levels are measured in 1st, 3rd and 5th postoperative day (POD). Patients' characteristics (age, sex, renal function, comorbidities), tumor localization, type of operation, intra and postoperative complications and their management, reinterventions, length of hospital stay are recorded. Inclusion criteria are: patients undergoing all different kinds of colorectal surgery (from right colectomies to low anterior resection), either in elective or emergent setting, either for cancer or benign disease (ex diverticular disease) with an anastomosis being performed (ileo-colic, colo-colic, or colo-rectal). Exclusion criteria are: age < 18 years, pregnant women, patients undergoing abdomino-perineal resection or other kinds of colorectal-surgery without an anastomosis being performed. A written informed consent is obtained from all patients. The study is approved by our institution's Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing all different kinds of colorectal surgery(from right colectomies to low anterior resection) in our institution, in elective setting, either for cancer or benign disease (ex diverticular disease) with an anastomosis being performed (ileo-colic, colo-colic, or colo-rectal

Exclusion Criteria:

* age < 18 years,
* pregnant women,
* patients undergoing abdomino-perineal resection or other kinds of colorectal-surgery without an anastomosis being performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing all different kinds of colorectal surgery (from right colectomies to low anterior resection), in elective setting, either for cancer or benign disease (ex diverticular disease) with an anastomosis being performed (ileo-colic, colo-colic, or colo-rectal)
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak | within the first 30 days after he operation

SECONDARY OUTCOMES:
Intra-abdominal infection | within 30 days from the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Andrea University Hospital, Rome, Italy

REFERENCES:
- [Derived] Giaccaglia V, Salvi PF, Antonelli MS, Nigri G, Pirozzi F, Casagranda B, Giacca M, Corcione F, de Manzini N, Balducci G, Ramacciato G. Procalcitonin Reveals Early Dehiscence in Colorectal Surgery: The PREDICS Study. Ann Surg. 2016 May;263(5):967-72. doi: 10.1097/SLA.0000000000001365. PMID 26528879